CLINICAL TRIAL: NCT00070590
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Efficacy, Safety and Tolerability of Bosentan in Patients With Interstitial Lung Disease Associated With Systemic Sclerosis
Brief Title: Efficacy and Safety of Oral Bosentan in Pulmonary Fibrosis Associated With Scleroderma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-052-330; BUILD 2
Record Dates: First submitted 2003-10-06; First posted 2003-10-08 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Fibrosis; Scleroderma, Systemic
Keywords: Scleroderma; Fibrosing alveolitis; Build; bosentan
MeSH Terms: conditions — Pulmonary Fibrosis; Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Bosentan

INTERVENTIONS:
Drug: Bosentan

SUMMARY:
Clinical and experimental studies suggest that bosentan could delay the progression of interstitial lung disease (ILD) associated with systemic sclerosis (SSc), a condition for which no established efficacious treatment is available. The present trial investigates a possible use of oral bosentan, which is currently approved for the treatment of symptoms of pulmonary arterial hypertension (PAH) WHO Class III and IV, to a new category of patients suffering from ILD associated with SSc.

ELIGIBILITY:
Main inclusion criteria:

* Systemic Sclerosis diffuse or limited
* Significant Interstitial Lung Disease on HRCTscan
* DLco < 80% predicted
* Dyspnea on exertion
* Walk not limited by musculoskeletal reasons

Main exclusion criteria:

* Interstitial Lung Disease due to other conditions than SSc
* End stage restrictive or obstructive lung disease
* Severe cardiac or renal diseases
* Significant pulmonary arterial hypertension
* Smoker (> 5cig./day)
* Treatment with immunosuppressive, antifibrotic drugs, high dose corticosteroids (within 4 weeks of randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2003-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to End-of-Study in 6-minute walk distance.

SECONDARY OUTCOMES:
Time to death (all causes) or to worsening of PFTs up to End-of-Study.
Worsening of PFTs (on 2 consecutive tests at least 4 weeks apart) is defined as: decrease from baseline ≥ 10% in FVC OR decrease from baseline ≥ 15% in DLco AND ≥ 6% in FVC

REFERENCES:
- [Derived] Liu C, Chen J, Gao Y, Deng B, Liu K. Endothelin receptor antagonists for pulmonary arterial hypertension. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD004434. doi: 10.1002/14651858.CD004434.pub6. PMID 33765691
- [Derived] Seibold JR, Denton CP, Furst DE, Guillevin L, Rubin LJ, Wells A, Matucci Cerinic M, Riemekasten G, Emery P, Chadha-Boreham H, Charef P, Roux S, Black CM. Randomized, prospective, placebo-controlled trial of bosentan in interstitial lung disease secondary to systemic sclerosis. Arthritis Rheum. 2010 Jul;62(7):2101-8. doi: 10.1002/art.27466. PMID 20506355